CLINICAL TRIAL: NCT05782855
Title: ROBot Assisted Physical Training of Older Patients During acUte hospitaliSaTion (ROBUST) - a Randomised Controlled Trial
Brief Title: ROBot Assisted Physical Training of Older Patients During acUte hospitaliSaTion
Acronym: ROBUST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Ryg, Professor, Consultant, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ROBUST
Record Dates: First submitted 2022-12-27; First posted 2023-03-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Functional Decline; ADL; Physical Inactivity; Acute Illness
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): Participants in the control group will receive usual individualized training with a physiotherapist and passive sham training of lower extremities with the rehabilitation robot twice a day until day of discharge. The physiotherapist will be blinded to allocation. Sham training consists of 3 sets of 8 passive repetitions with each leg twice a day.
  Interventions: Other: Passive Robot assisted physical training during acute hospitalisation
- Intervention group (Active Comparator): The intervention group will receive usual individualized training with a physiotherapist and active strength training of lower extremities by the robot twice a day until day of discharge. The physiotherapist will be blinded to allocation. Training will focus on the muscle groups in the lower extremities, which are used to get up from a chair and walk around (thigh- and calf muscles). Active training consists of 3 sets of maximum repetitions with a minimum of 65% (65-80%) intensity of 1 RM with each leg twice a day.
  Interventions: Other: Active Robot assisted physical training during acute hospitalisation

INTERVENTIONS:
Other: Active Robot assisted physical training during acute hospitalisation — Active training is delivered by an innovative training robot (ROBERT®). The robot is handled by staff who attaches the robot to the patient's leg. The staff programs the exercise movement, whereby the robot remembers the movement. The robot holds the patient's leg and perform extension of hip and knee. The patient must use their muscular power to stretch the leg while ROBERT® provides resistance.
  Training is defined as a minimum of three sessions before discharge.
  Arms: Intervention group
Other: Passive Robot assisted physical training during acute hospitalisation — Passive training is delivered by an innovative training robot (ROBERT®). The robot is handled by staff who attaches the robot to the patient's leg. The staff programs the movement, whereby the robot remembers the movement. The robot holds the patient's leg and perform passive extension of hip and knee. ROBERT® moves the leg independently without the patient using any muscle power.
  Training is defined as a minimum of three sessions before discharge.
  Arms: Control group

SUMMARY:
This study aims to address if robot assisted physical training can prevent functional decline during acute hospitalisation in older geriatric patients.

Design: blinded RCT. Patients: n = 488. Primary outcome is functional decline, assessed by Barthel-Index and 30s chair stand test. One- and three months follow-up.

DETAILED DESCRIPTION:
Introduction:

Inactivity during hospitalisation is associated with significant risk of functional decline especially in older patients. This have major impact on the individual level due to decreased wellbeing and higher level of dependency and on the society level due to increased caregiver burden following hospital discharge. This study aims to address if robot assisted physical training can prevent functional decline during acute hospitalisation in older geriatric patients.

Methods:

ROBUST is a blinded RCT. Patients (n = 488) admitted with acute medical illness to Department of Geriatric Medicine, Odense University Hospital will be randomised to usual care and robot assisted active strength training of lower extremities twice daily (intervention group) or usual care and robot assisted passive sham training (control group) until discharge. Both groups will receive protein supplements.

Inclusion criteria: ≥65 years of age, able to ambulate before hospitalisation, expected length of stay ≥2 days.

Exclusion criteria: Able to ambulate without assistance during current hospitalisation, severe dementia, delirium, conditions contradicting robot training.

The primary outcome, functional decline, will be assessed by Barthel-Index and 30s chair stand test.

Secondary outcomes include Quality of life (EQ-5D), Geriatric Depression Scale, Fear of falling (FES-I), cognition (MMSE), qualitative interviews, falls, caregiver burden, discharge destination, readmissions, healthcare costs, sarcopenia, and mortality.

Outcomes will be assessed at admission, discharge, and one- and three months follow-up. Data on comorbidity, medications, blood samples, and clinical frailty scale will be collected.

Discussion: This study will investigate the effects of in-hospital robot assisted strength training on functional status in older patients with multimorbidity.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* Able to ambulate before hospitalisation (with/without assistance)
* Able to communicate with the research team
* Expected length of stay ≥2 days
* Residing on Funen, Denmark

Exclusion Criteria:

* Able to ambulate without assistance during current hospitalisation
* Known severe dementia
* Positive Confusion and Assessment Method score (20)
* Patients who have received less than 3 training sessions at discharge
* Terminal illness
* Recent major surgery or lower extremity bone fracture in the last 3 months
* Conditions contradicting use of ROBERT (unstable vertebral-, pelvic, or lower extremity fractures; high intracranial pressure; pressure ulcers or risk of developing pressure ulcers due to fragile skin; patients with medical instability)
* Metastases at femur or hip
* Deemed not suitable for mobilization sessions with the robot by the healthcare professional
* If the patient weighs more than 165 kg (the robot cannot lift the leg if the patient is severely overweight)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Barthel Index 100 | Change from baseline (day of hospital admission) to day of hospital discharge (an average of 1 week)
  Functional evaluation assessed by Barthel Index 100. The Barthel Index is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.
Change from baseline 30 Second Sit to Stand Test | Change from baseline (day of hospital admission) to day of hospital discharge (an average of 1 week)
  Functional evaluation assessed by 30 Second Sit to Stand Test . The 30 Second Sit to Stand Test is for testing leg strength and endurance in older adults.

SECONDARY OUTCOMES:
Quality of life EQ-5D | Day of hospital admission; day of hospital discharge (an average of 1 week); 1 month follow-up; 3 months follow-up.
  Quality of life is assessed using the questionaire Quality of life EuroQol-5 dimension (EQ-5D). The EQ-5D comprises five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) each with three levels (no problems, some problems, extreme problems/unable), thus generating 243 possible health states.
  The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Mood status | Day of hospital admission; day of hospital discharge (an average of 1 week); 1 month follow-up; 3 months follow-up.
  Mood status are assessed by the 15-item Geriatric Depression Scale. The Short Form GDS consisting of 15 questions. Of the 15 items, 10 indicated the presence of depression when answered positively, while the rest indicated depression when answered negatively. Scores of 0-4 are considered normal, depending on age, education, and complaints; 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Concern about falling including number of falls | Day of hospital admission; day of hospital discharge (an average of 1 week); 1 month follow-up; 3 months follow-up.
  Concern about falling is assessed using the 16-item Short Falls Efficacy Scale International (Short FES-I) questionaire. To calculate the Short FES-I score when all items are completed, simply add the scores for each item together to give a total that ranges as follows: minimum 7 (no concern about falling) to maximum 28 (severe concern about falling).
Patient perspective by qualitative interviews | Day of hospital discharge (an average of 1 week); 1 month follow-up.
  Qualitative semi-structured in-depth interviews will be performed with at least 12 patients at discharge and 1 month follow-up to explore their perspectives and experiences (PRO/PRE). The qualitative interviews will provide further and deeper explanations of the results from the quantitative parts of the study. By using this mixed-methods approach the research results will be strengthen by the complementary findings. The analysis of the qualitative data will be completed in line with manifest content analysis by Graneheim and Lundman. Data will be handled using the software NVivo
Cognitive function | Day of hospital admission; day of hospital discharge (an average of 1 week); 1 month follow-up; 3 months follow-up.
  Cognitive function is assessed by the Mini Mental State Examination. The Mini-Mental State Examination (MMSE) is a set of 11 questions that is used to check for cognitive impairment (problems with thinking, communication, understanding and memory). The maximum score for the MMSE is 30. A score of 25 or higher is classed as normal. If the score is below 24, the result is usually considered to be abnormal, indicating possible cognitive impairment.
Muscle quantity | Day of hospital admission; day of hospital discharge (an average of 1 week); 1 month follow-up; 3 months follow-up.
  Muscle quantity is assessed using bioelectrical impedance by InBodyS10. Bioelectrical impedance analysis (BIA) is a method for estimating body composition, in particular body fat and muscle mass.
Sarcopenia | Day of hospital admission; day of hospital discharge (an average of 1 week); 1 month follow-up; 3 months follow-up.
  Sarcopenia is assessed based on the 2019 European guidelines by Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyère O, Cederholm T, et al.
Need of care at home | From 3 months prior to day of hospital admission to 3 months following day of hospital discharge.
  Individual level data from the municipalities will be used to assess amount of need of care/home care provided by the municipality 3 months before admission and 3 months after discharge. Need of care at home is devided in the following categories: practical help, personnel care, nursing and training. Amount of need of care will be presented in hours.
Length of hospital stay | From day of hospital admission to day of hospital discharge (an average of 1 week).
  Length of hospital stay will be defined as number of days in geriatric department.
Discharge destination | Day of hospital discharge (an average of 1 week).
  Data about discharge destination will be collected at the day of discharge (own home, temporary rehabilitation units, nursing homes)
Rate of hospital readmission | 30 days following day of hospital discharge.
  Patients will be followed through a review of medical records for any unplanned hospitalisation within 1 month after discharge.
  Readmission definition: any unplanned hospital contact with a duration of 12+hours, occurring between 4 hours and 30 days after discharge from the Department of Geriatric Medicine.
Health care cost evaluation | 3 months follow-up.
  A researcher in health care economics will perform a health care cost evaluation addressing running cost using ROBERT, discharge destination, hospital readmissions, care giver burden, and visits to the general practitioner after 3 months.
Mortality | 1- and 3-months follow-up.
  Administrative registers will be used to assess mortality at 1- and 3- months follow-up.
Change from baseline Barthel Index 100 | Change from baseline (day of hospital admission) to 1 month follow-up and 3 months follow-up.
  Functional evaluation assessed by Barthel Index 100. The Barthel Index is an ordinal scale used to measure performance in activities of daily living (ADL). Ten variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.
Change from baseline 30 Second Sit to Stand Test | Change from baseline (day of hospital admission) to 1 month follow-up and 3 months follow-up.
  Functional evaluation assessed by 30 Second Sit to Stand Test . The 30 Second Sit to Stand Test is for testing leg strength and endurance in older adults.
Clinical Frailty Scale | Change from baseline (day of hospital admission) to 1 month follow-up and 3 months follow-up.
  The 9-point Clinical Frailty Scale (CFS) with pictograms is used at baseline before randomisation, at discharge, and at 1- and 3-month follow-up (28) to examine the impact of the exercise intervention on frailty and to determine the impact of baseline frailty on the effectiveness of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Ryg, Professor, Principal Investigator — Department of geriatric medicine Odense University hospital, Denmark
Locations (1):
- Odense University Hospital/Svendborg Hospital, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bertelsen AS, Storm A, Minet L, Ryg J. Use of robot technology in passive mobilization of acute hospitalized geriatric medicine patients: a pilot test and feasibility study. Pilot Feasibility Stud. 2020 Jan 6;6:1. doi: 10.1186/s40814-019-0545-z. eCollection 2020. PMID 31921434
- [Derived] Bertelsen AS, Masud T, Suetta C, Rosenbek Minet L, Andersen S, Lauridsen JT, Ryg J. ROBot-assisted physical training of older patients during acUte hospitaliSaTion-study protocol for a randomised controlled trial (ROBUST). Trials. 2024 Apr 4;25(1):235. doi: 10.1186/s13063-024-08044-6. PMID 38576046

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT05782855/SAP_001.pdf